CLINICAL TRIAL: NCT02771483
Title: Giant Cell Arteritis and PET Scan (GAPS) Study - Improving the Diagnosis and Prognostication of Giant Cell Arteritis Through the Novel Use of Positron Emission Tomography and Immune Biomarkers
Brief Title: Giant Cell Arteritis and PET Scan (GAPS) Study
Status: Completed | Type: Observational
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Anthony Sammel, Rheumatology fellow, Royal North Shore Hospital
Other Study IDs: RESP/16/44
Record Dates: First submitted 2016-05-09; First posted 2016-05-13 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Temporal artery specimens Serology
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Suspected GCA (GCA final diagnosis)
- Suspected GCA (alternative final diagnosis)

SUMMARY:
Giant cell arteritis (GCA) is a medium to large vessel vasculitis with a predilection for the superficial cranial and intrathoracic arteries. Diagnosing the condition and predicting which patients will develop large vessel complications remains a challenge. There are limitations with temporal artery biopsy, magnetic resonance angiography and ultrasound of temporal arteries and American College of Rheumatology classification criteria.

Positron emission tomography (PET) has been shown to be a useful modality in detecting inflammation in large intra-thoracic vessels but previously has not been able to accurately detect FDG uptake in the superficial cranial arteries due to poor spatial resolution. Newer scanners can perform finer cuts of the head and can detect uptake in these arteries.

This study has three main components:

1. Cross sectional study assessing the accuracy of PET uptake in the superficial cranial and intrathoracic arteries of suspected GCA patients for the diagnosis of GCA
2. Cohort study assessing the prognostic implication of FDG aortic uptake on aortic diameter at 24 months
3. Cohort study assessing the Th1 and Th17 cytokine profile in patients with and without FDG PET uptake at 0, 6 and 24 months

ELIGIBILITY:
Inclusion Criteria:

* Rheumatologist, neurologist or ophthalmologist suspect diagnosis of GCA
* Age > 50
* Meet at least 2 of 1990 American College of Rheumatology classification criteria for GCA

  1. Age >= 50
  2. ESR >= 50
  3. New onset localised headache
  4. Temporal artery abnormality (tenderness or decreased pulsation)
  5. Positive biopsy (will not be available at time of enrolment)

Exclusion Criteria:

* Corticosteroid therapy for > 72 hours before first PET scan
* Prolonged corticosteroid therapy (> 1 week) for another indication in past 6 months
* History of vasculitis or connective tissue disease
* Active malignancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected GCA
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of FDG uptake in the superficial cranial or intrathoracic arteries for the diagnosis of temporal artery biopsy proven GCA amongst patients with suspected GCA | Baseline

SECONDARY OUTCOMES:
Difference in aortic diameter at 24 months between patients with and without PET scan aortic uptake at time 0. | 24 months
Difference in Th1 and Th17 axis cytokines in patients with and without thoracic large vessel PET uptake at 0, 6 and 24 months | 24 months
Prevalence of varicella zoster virus antigen and DNA in temporal artery biopsy GCA specimens | 24 months
Prevalence of acute varicella zoster IgM serology positivity in biopsy confirmed GCA patients | 24 months
Difference in combined vascular events between GCA patients with and without thoracic large vessel PET uptake at 0, 6 and 24 months | 24 months
Difference in temporal artery histology between GCA patients with and without thoracic large vessel PET uptake at 0 months | Baseline
Difference in temporal artery histology between GCA patients with and without temporal artery PET uptake at 0 months | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Anthony M Sammel, MBBS, Principal Investigator — Royal North Shore Hospital, St Leonards, Australia
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sammel AM, Hsiao E, Schembri G, Nguyen K, Brewer J, Schrieber L, Janssen B, Youssef P, Fraser CL, Bailey E, Bailey DL, Roach P, Laurent R. Diagnostic Accuracy of Positron Emission Tomography/Computed Tomography of the Head, Neck, and Chest for Giant Cell Arteritis: A Prospective, Double-Blind, Cross-Sectional Study. Arthritis Rheumatol. 2019 Aug;71(8):1319-1328. doi: 10.1002/art.40864. Epub 2019 Jun 12. PMID 30848549